CLINICAL TRIAL: NCT04268576
Title: Impact of an Improved Rehabilitation Program After a Scheduled Hysterectomy.
Acronym: RAACHYS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-08-CHRMT
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Post-Op Complication
Keywords: hysterectomy; post operative
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is an observational study, prospective in order to assess the impact of the implementation of an early rehabilitation program on post-operative recovery. this is measured by the qOR15 questionnaire in patients operated on for a programmed hysterectomy, it takes place in the gynecology department of the CHR Metz-Thionville hospital.

DETAILED DESCRIPTION:
This program implemented will comply with HAS recommendations. The only change in management for patients participating in the study is the completion of the self-questionnaire QOR-15 on D-1 (the day before surgery), D0 (the day of the surgery) and D1 (the day after the surgery).

It is planned to include 74 patients before the implementation of the early rehabilitation protocol and 74 patients after the implementation of the early rehabilitation protocol. The total duration of inclusion is established at 18 months.

The measures applied should improve the patient's well-being and accelerate his return to normal life and therefore reduce the length of his stay.

ELIGIBILITY:
Inclusion Criteria:

* Indication of a scheduled hysterectomy
* Presence of a utero-ovarian affection, deemed resectable and requiring a regulated hysterectomy (outside the context of the emergency) associated or not with pelvic or lumbar-aortic dissection.
* classified ASA 1 to 3
* informed about the principles of improved rehabilitation by the surgeon and the anesthesiologist + written document (accessible on the site www.grace-asso.fr).
* able to return home after discharge from the hospital, having a telephone and being able to contact their doctor or the service if necessary or transferred to a convalescent home at their request.

Exclusion Criteria:

* Patients included in another study
* Refusal to use data by the patient
* Inability to respond to self-questionnaires due to cognitive impairment, difficulties in reading or understanding the French language
* Patients included in another study
* Patients with severe or unbalanced associated conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected according to the inclusion and exclusion criteria when they go to the operating room. It is planned to include 74 patients for rehabilitation before the implementation of the protocol and 74 patients after the implementation of the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the QoR-15 score D1 | day 1
  The QoR score 15 is a self-questionnaire of 15 items, each scored from 0 to 10. These items assess 5 dimensions of post-operative recovery: pain, physical comfort, functional autonomy, emotions and psychological support. These 15 items represent the quality of post-operative rehabilitation in its physical and mental dimensions.
  A variation of 8 points is considered significant.

SECONDARY OUTCOMES:
Overall duration of the hospital stay D-1 | One day before surgery
  Overall duration of the hospital stay in days
Overall duration of the hospital stay day of discharge from hospital | Up to 30 days
  Overall duration of the hospital stay in days
Duration of fasting pre and post-operative | Up to 30 days
  Duration of fasting pre and post-operative in hours
Post-operative nausea / vomiting Day 0 | Day of surgery
  Occurrence of nausea / vomiting postoperative (yes / no)
Post-operative nausea / vomiting D+1 | One day after surgery
  Occurrence of nausea / vomiting postoperative (yes / no)
Post-operative nausea / vomiting day of hospital discharge | Up to 30 days
  Occurrence of nausea / vomiting postoperative (yes / no)
Intraoperative maximum Visual Analog Scale (VAS) on day 0 | day 0
  Maximum Visual Analog Scale (VAS) (from 0 to 100mm), 0 mm (minimum, none) 100 mm (maximum, worst pain possible)
Intraoperative maximum visual analog scale (VAS) on day 1 | One day after surgery
  Maximum Visual Analog Scale (VAS) (from 0 to 100mm), 0 mm (minimum, none) 100 mm (maximum, worst pain possible)
Intraoperative maximum visual analog scale (VAS) on day of discharge from hospital | Up to 30 days
  Maximum Visual Analog Scale (VAS) (from 0 to 100mm), 0 mm (minimum, none) 100 mm (maximum, worst pain possible)
Time to return gastrointestinal function | Up to 30 days
  Transit recovery time in hours
Enhancement of gastrointestinal motility on Day 0 | day 0
  Whether or not chewing gum is taken (yes/no)
Enhancement of gastrointestinal motility on day 1 | One day after surgery
  whether or not chewing gum is taken (yes/no)
Enhancement of gastrointestinal motility on the day of discharge from the hospital | Up to 30 days
  whether or not chewing gum is taken (yes/no)
Presence of a urinary catheter or drain in postoperative | day 0
  Presence of a urinary catheter or drain in postoperative (yes / no)
Time before first standing | Up to 30 days
  Time before first standing in hours
occurrence of postoperative complications | day 30
  occurrence of postoperative complications (resumption of surgery at 30 days)
Evaluation of the QoR-15 score D0 | Day 0
  The QoR score 15 is a self-questionnaire of 15 items, each scored from 0 to 10. These items assess 5 dimensions of post-operative recovery: pain, physical comfort, functional autonomy, emotions and psychological support. These 15 items represent the quality of post-operative rehabilitation in its physical and mental dimensions.
  A variation of 8 points is considered significant.
Evaluation of the QoR-15 score D-1 | Day -1
  The QoR score 15 is a self-questionnaire of 15 items, each scored from 0 to 10. These items assess 5 dimensions of post-operative recovery: pain, physical comfort, functional autonomy, emotions and psychological support. These 15 items represent the quality of post-operative rehabilitation in its physical and mental dimensions.
  A variation of 8 points is considered significant.
Rate of laparotomy | day 0
  percentage
Mobility on day 0 | day 0
  The time between the end of surgery and the first time to get up in hours,
Mobility on day 1 | One day after surgery
  The time between the end of surgery and the first time to get up in hours
Mobility on the day of discharge from the hospital | Up to 30 days
  The time between the end of surgery and the first time to get up in hours

CONTACTS AND LOCATIONS:
Overall Officials: Antoine BECRET, MD, Principal Investigator — CHR Metz-Thionville
Locations (1):
- CHR Metz-Thionville, Metz, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin F, Vautrin N, Elnar AA, Goetz C, Becret A. Evaluation of the impact of an enhanced recovery after surgery (ERAS) programme on the quality of recovery in patients undergoing a scheduled hysterectomy: a prospective single-centre before-after study protocol (RAACHYS study). BMJ Open. 2022 Apr 7;12(4):e055822. doi: 10.1136/bmjopen-2021-055822. PMID 35393312